CLINICAL TRIAL: NCT06160557
Title: A Single-arm, Prospective, Multi-center Phase II Clinical Study of Non-curative Resection Plus Radiotherapy After Endoscopic ESD for Superficial Esophageal Squamous Cell Carcinoma
Brief Title: A Clinical Study of Non-curative Resection Plus Radiotherapy After Endoscopic ESD for Superficial Esophageal Squamous Cell Carcinoma
Status: Enrolling by invitation | Type: Observational
Sponsor: Xiaomeng Zheng (Other)
Responsible Party: Sponsor-Investigator, Xiaomeng Zheng, Master Degree Candidate, Fujian Medical University
Organization: Fujian Medical University (Other)
Other Study IDs: non-curative ESD
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Esophagus Cancer; Radiotherapy; Endoscopic Mucosal Resection
Keywords: esophageal squamous carcinoma; Radiotherapy; endoscopic submucosal dissection
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of observational study is to learn about the outcomes of the participants. The main questions it aims to answer are:

1. ESD additional postoperative radiotherapy in patients with non healing SESCC overall survival (OS) and disease-free survival (DFS)
2. The adverse events (AE) of additional radiotherapy after ESD for non-curative SESCC patients were counted, and its safety was evaluated.

Participants will receive radiation therapy as necessary.

DETAILED DESCRIPTION:
This study is an in ESD subjects, early postoperative esophageal cancer pathology returns have cut edge positive, lymphatic vascular invasion, SM2 - SM3 or pathologic stage under the condition of low degree of differentiation, observe additional radiation noninferiority and safety of single arm, multicenter, phase II clinical study.

The test plan into the group of 40 cases of the subjects, the ESD additional postoperative radiotherapy group, using three dimensional conformal radiation therapy and intensity-modulated radiation therapy technology. Good ESD within 2 months, after the ulcer healing began RT as a supplementary treatment. All patients underwent CT simulation before treatment, and the location of the tumor bed was determined according to the lesion location under ultrasound gastroscopy before ESD and the scar tissue formed after ESD. If necessary, titanium clips were placed under gastroscopy before the first radiotherapy to locate the tumor bed, that is, GTVtb. CTV1 of cervical and middle and upper thoracic esophageal cancer included bilateral supraclavicular and mediastinal lymph nodes to the tracheal bifurcation area, the so-called "short T" field. CTV1 of lower thoracic esophageal cancer includes mediastinum, perigastric and lymphatic drainage areas above the celiac trunk. Plans to target (PTV) has CTV1 outside enlarge margins of 0.5 cm. The dose to PTV was 45Gy/25 fractions /5 weeks (5 days/week), and the dose to PGTVtb was 50Gy/25F(simultaneous boost). For patients with positive margins, the PTV dose was 48Gy/30 fractions /6 weeks (5 days/week), and the PGTVtb dose was 60Gy/30 fractions. The study was followed up for a total of 3 years. During the study period, the subjects were evaluated by tumor imaging before and after the additional radiotherapy. All participants were treated until disease progression, development of unacceptable toxicity, receipt of new antineoplastic therapy, withdrawal of informed consent, loss to follow-up, or death, or other conditions judged by the investigator to warrant discontinuation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* (1) patients with esophageal squamous cell carcinoma within pT1 (stage pT1N0M0) confirmed by pathology;
* (2) The following conditions were confirmed by pathology after ESD: submucosal invasion > 200μm (stage SM2-SM3), undifferentiated or poorly differentiated pathological degree, positive surgical margin, vascular and lymphatic invasion;
* (3) aged 18-75 years old (inclusive);
* (4) predicted survival time ≥6 months;
* (5) ECOG score of 0-1;
* (6) no obvious other symptoms or no effect assessed by researchers;
* (7) Women of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose. Male or female patients of childbearing potential volunteered to use an effective contraceptive method, such as dual barrier methods, condoms, oral or injectable contraceptives, intrauterine devices, etc., during the study and for 90 days after the last study medication was taken. All female patients will be considered fertile unless the woman has undergone natural menopause, artificial menopause, or sterilization (e.g., hysterectomy, bilateral adnexectomy);
* (8) Electrocardiogram, blood, biochemical and other basic examinations had no contraindications to radiotherapy, and had sufficient bone marrow, liver and kidney organ functions. Laboratory examinations within 7 days before the first dose of medication met the following requirements: a. Absolute neutrophil count (ANC) ≥1.5×109/L, platelet ≥100×109/L and hemoglobin ≥90g/L (no blood transfusion, blood products, granulocyte colony-stimulating factor or other hematopoietic stimulating factor correction within 14 days before laboratory tests); b. Serum total bilirubin ≤1.5 times the upper limit of the normal reference range (× ULN); c. alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5 × ULN; d. Serum creatinine ≤1.5 × ULN and creatinine clearance ≥50 mL/min, (calculated by Cockcroft/Gault formula) : Female: Ccr= (140-age) x weight (kg) x 0.85/(72 x serum creatinine (mg/dL)) Male: Ccr= (140-age) x body weight (kg) x 1.00 /(72 x serum creatinine (mg/dL)); e. Urine routine examination showed urine protein < 2+; If urinary protein is ≥2+, 24-hour urinary protein should be less than 1 g; f. Sufficient coagulation function, international normalized ratio (INR) ≤1.5, prothrombin time (PT), activated partial prothrombin time (APTT) ≤1.5 × ULN; If the subject is receiving anticoagulant therapy, as long as the PT is within the prescribed range of anticoagulant drugs;
* (9) patients who know all available treatment options and understand the advantages and disadvantages of each option and are willing to enroll after being fully informed;
* (10) consent to provide tissue examination specimens for further confirmation of pathological grade if necessary;
* (11) Suitability for inclusion in the study was determined by two physicians with senior professional titles or above independently;
* (12) have fully understood and voluntarily provided informed consent for the study (prior to any trial-specified procedures) and be able to comply with protocol-specified visits and related procedures.

Exclusion Criteria:

* (1) growth period on contraception, pregnancy (test positive for drug use before pregnancy) or lactating women;
* (2) patients currently have any disease or condition affect drug absorption, or patients cannot oral medicine;
* (3) patients with other malignant tumors (except well-controlled basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, non-melanoma skin cancer, or lentigo malignant nevus) within the past 5 years or with concurrent systemic malignant tumors;
* (4) Patients with other chronic diseases had contraindications to radiotherapy;
* (5) the presence of any active autoimmune disease requiring systemic treatment or a history of autoimmune disease within the past 2 years, including but not limited to interstitial pneumonia, uveitis, inflammatory bowel disease, hepatitis, hypophysitis, vasculitis, systemic lupus erythematosus, etc. (vitiligo, psoriasis, alopecia, or Graves' disease without systemic treatment within the past 2 years; Only need insulin replacement therapy of patients with type 1 diabetes can be incorporated into); Known primary immunodeficiency disease; For patients with only positive autoimmune antibodies, the presence of autoimmune diseases should be determined according to the investigator's judgment;
* (6) receiving systemic immunostimulant therapy within 4 weeks before the first dose;
* (7) administration of any live or live attenuated vaccine within 4 weeks before the first dose or planned during the study period;
* (8) patients who underwent major surgery (the definition of major surgery referred to grade 3 and grade 4 surgery specified in the "Administrative Measures for the Clinical Application of Medical Technology" implemented on May 1, 2009) or unhealed wounds, ulcers or fractures within 4 weeks before the first medication;
* (9) Patients had drug-uncontrolled hypertension defined as systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg;
* (10) patients with active gastric and duodenal ulcer, ulcerative colitis and other gastrointestinal diseases, or unresected tumors with active bleeding, or other conditions that may cause gastrointestinal bleeding or perforation as judged by the investigators;
* (11) for the first time 2 months before using this drug has a history of thrombosis or bleeding tendency obviously evidence or patients (> 30 mL, 2 months bleeding appear hematemesis, black dung, bloody), haemoptysis > 5 mL (4 weeks) of fresh blood, PICC except caused by blood clots;
* (12) for the first time happened within six months before using this drug arterial thrombosis or deep vein thrombosis; Or had a stroke event and/or transient ischemic attack within 12 months;
* (13) clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting within 6 months before the first dose of medication; Congestive heart failure (New York heart association (NYHA) class 2 or higher. Left ventricular ejection fraction (LVEF) <50%;
* (14) any arterial thromboembolic event, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, occurred within 6 months before enrollment;
* (15) History of deep vein thrombosis, pulmonary embolism, or any other major thromboembolism within 3 months before enrollment (superficial venous thrombosis was not considered a "major" thromboembolism);
* (16) patients with active tuberculosis (TB), is receiving anti-tuberculosis treatment or medication for the first time 1 year before received anti-tuberculosis treatment;
* (17) patients with previous or current history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severe impaired pulmonary function, etc.;
* (18) the known history of allogeneic organ transplantation and the history of allogeneic hematopoietic stem cell transplantation;
* (19) patients with active infection occurred prior to or during the screening, first radiotherapy fever of unknown origin (temperature > 38.5 oC);
* (20) clinically significant severe electrolyte abnormalities as judged by the investigator;
* (21) significant malnutrition, such as need intravenous supplement nutrient solution; The exception was correction of malnutrition for more than 4 weeks before the first treatment;
* (22) The patient had uncured hyperthyroidism;
* (23) other acute or chronic medical conditions, psychiatric conditions, or abnormal laboratory values that could increase the risk associated with the study treatment or interfere with the interpretation of the study results and would, in the investigator's judgment, have made the patient ineligible for the study;
* (24) uncontrolled metabolic disorders or other non-malignant organ or systemic diseases or secondary effects of cancer, and may lead to high medical risk and/or uncertainty in the evaluation of survival;
* (25) The investigator considered that the patient was not suitable to participate in the study for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among the patients with early esophageal cancer after ESD, the pathological results showed positive surgical margin, lymphovascular invasion, SM2-SM3 stage, or poor pathological differentiation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival, OS | It continued for 3 years after enrollment
  OS is defined as the interval from the date of enrollment to the death of the subject from any cause.
Disease Free Survival, DFS | It continued for 3 years after enrollment
  DFS is defined as the interval from the date of enrollment to first disease progression, whichever occurred first.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China